CLINICAL TRIAL: NCT01018641
Title: A Phase 1 Trial To Evaluate The Safety, Tolerability, And Immunogenicity Of 3 Ascending Dose Levels Of A 3-Antigen Staphylococcus Aureus Vaccine (SA3Ag) In Healthy Adults
Brief Title: An Evaluation Of Three Dose Levels Of 3-Antigen Staphylococcus Aureus Vaccine (SA3Ag) In Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 6123K1-1007; B2251002
Record Dates: First submitted 2009-11-20; First posted 2009-11-23 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Bacterial Infections; Staphylococcal Vaccines; Immunotherapy, Active; Staphylococcal Skin Infections; Staphylococcal Infections
Keywords: Staphylococcus aureus; Vaccine
MeSH Terms: conditions — Bacterial Infections; Motor Activity; Staphylococcal Skin Infections; Staphylococcal Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental): SA3Ag in both stage 1 and stage 2
  Interventions: Biological: SA3Ag vaccine; Procedure: Blood draw; Procedure: Colonization swab samples
- 2 (Experimental): SA3Ag in stage 1 followed by placebo in stage 2.
  Interventions: Biological: SA3Ag followed by Placebo; Procedure: Blood draw; Procedure: Colonization swab samples
- 3 (Placebo Comparator): Placebo in both stage 1 and stage 2
  Interventions: Biological: Placebo; Procedure: Blood draw; Procedure: Colonization swab samples
- 4 (Experimental): SA3Ag in stage 1 and no vaccine in stage 2.
  Interventions: Biological: SA3Ag with no booster in stage 2; Procedure: Blood draw; Procedure: Colonization swab samples
- 5 (Placebo Comparator): Placebo in stage 1 and no vaccine in stage 2.
  Interventions: Procedure: Placebo with no booster in stage 2; Procedure: Blood draw; Procedure: Colonization swab samples

INTERVENTIONS:
Biological: SA3Ag vaccine — In stage 1, each subject will receive 1 injection (0.5 mL) of one of the following doses:
  Low dose level 10 μg of CP5 and CP8 and 20 μg of rClfAm Mid-dose level 30 μg of CP5 and CP8 and 60 μg of rClfAm High dose level 100 μg of CP5 and CP8 and 200 μg of rClfAm
  In stage 2 the subject will receive 0.5 mL IM of the same dose level he/she received in stage 1.
  Arms: 1
Procedure: Blood draw — Blood for immunogenicity will be taken at timepoints throughout stage 1 and stage 2. Blood for hematology will be done in a select subset of subjects in stage 1.
  Arms: 1
Procedure: Colonization swab samples — Colonization swabs will be taken at timepoints throughout stage 1 and stage 2.
  Arms: 1
Biological: SA3Ag followed by Placebo — In stage 1, each subject will receive 1 injection (0.5 mL) of one of the following doses:
  Low dose level 10 μg of CP5 and CP8 and 20 μg of rClfAm Mid-dose level 30 μg of CP5 and CP8 and 60 μg of rClfAm High dose level 100 μg of CP5 and CP8 and 200 μg of rClfAm
  In stage 2 the subject will receive one injection of 0.5 mL IM of the placebo.
  Arms: 2
Procedure: Blood draw — Blood for immunogenicity will be taken at timepoints throughout stage 1 and stage 2. Blood for hematology will be done in a select subset of subjects in stage 1.
  Arms: 2
Procedure: Colonization swab samples — Colonization swabs will be taken at timepoints throughout stage 1 and stage 2.
  Arms: 2
Biological: Placebo — In both stage 1 and stage 2, recipients will receive one injection (0.5 mL) IM of 150 mM (isotonic) NaCl for a total of 2 injections throughout the study.
  Arms: 3
Procedure: Blood draw — Blood for immunogenicity will be taken at timepoints throughout stage 1 and stage 2. Blood for hematology will be done in a select subset of subjects in stage 1.
  Arms: 3
Procedure: Colonization swab samples — Colonization swabs will be taken at timepoints throughout stage 1 and stage 2.
  Arms: 3
Biological: SA3Ag with no booster in stage 2 — In stage 1, each subject will receive 1 injection (0.5 mL) of one of the following doses:
  Low dose level 10 μg of CP5 and CP8 and 20 μg of rClfAm Mid-dose level 30 μg of CP5 and CP8 and 60 μg of rClfAm High dose level 100 μg of CP5 and CP8 and 200 μg of rClfAm
  In stage 2 the subject will receive no vaccine.
  Arms: 4
Procedure: Blood draw — Blood for immunogenicity will be taken at timepoints throughout stage 1 and stage 2. Blood for hematology will be done in a select subset of subjects in stage 1.
  Arms: 4
Procedure: Colonization swab samples — Colonization swabs will be taken at timepoints throughout stage 1 and stage 2.
  Arms: 4
Procedure: Placebo with no booster in stage 2 — In stage 1, recipients will receive one injection (0.5 mL) IM of 150 mM (isotonic) NaCl.
  In stage 2 the subject will receive no vaccine.
  Arms: 5
Procedure: Blood draw — Blood for immunogenicity will be taken at timepoints throughout stage 1 and stage 2. Blood for hematology will be done in a select subset of subjects in stage 1.
  Arms: 5
Procedure: Colonization swab samples — Colonization swabs will be taken at timepoints throughout stage 1 and stage 2.
  Arms: 5

SUMMARY:
This study is a first-in-human (Phase 1) study using three dose levels of an investigational vaccine directed against Staphylococcus aureus (SA3Ag). This study is primarily designed to assess how safe and well tolerated SA3Ag is, but will also describe the immune response over 12 months elicited by SA3Ag. Additionally, this study will assess the effect of SA3Ag vaccine on the number of Staphylococcus aureus bacteria that naturally occur on the skin and within the nose and throat.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 24 years or 50 to 85 years who are available for the entire duration of the study, able to be contacted by phone, and able to complete all study procedures, including completion of an electronic diary (e-diary).
* Men and women who are able to have children, must use a reliable method of birth control for the duration of the study.

Exclusion Criteria:

* Any major illness that would substantially increase the risk associated with participation in the study, or interfere with the evaluation of the study objectives - this is determined by the local physician.
* Donation of 250 mL or more of blood within the last 3 months.
* Condition associated with prolonged bleeding time, including subjects taking anticoagulant medication or antiplatelet therapy.
* Any contraindication to vaccination or vaccine components.
* Immunocompromised persons and subjects who receive treatment with immunosuppressive therapy.
* Previous administration of S. aureus vaccination.
* Receipt of blood products or immunoglobulins within 12 months prior to study
* Participation in another trial (not including observational trials) within the last 30 days.
* Study site personnel or immediate family members (first-degree relatives).
* Women who are pregnant (as determined by urine pregnancy test) or breast-feeding.
* Residence in a nursing home or long-term care facility or requirement for semiskilled nursing care.
* For subjects aged 65 years or older, a Mini-Mental State Examination (MMSE) score of <=21.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The primary immunogenicity endpoint in stage 1 is antigen-specific antibody levels using an Ig binding assay (Ig titers) 28 days after vaccination at visit 1 in the 50- to 85-year age stratum at each vaccine group (3 SA3Ag dose levels and placebo). | 1 month
The primary comparison of interest is a 2-fold increase in Ig titers relative to baseline for each antigen. | 1 month

SECONDARY OUTCOMES:
The secondary immunogenicity endpoints are Ig titers for each antigen (CP5, CP8, and rClfAm) 28 days after vaccination in the 18- to 24-year age stratum at each dose level cohort. | 1 month
Ig titers for each antigen 28 days after the booster dose. | 7 months
The safety endpoints are solicited and unsolicited AEs, SAEs, and hematologic and urine parameters. | 12 months
OPA titers for each antigen 28 days after vaccination in both age strata at selected dose level cohort(s). | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- Australia (5):
  - Pfizer Investigational Site, Herston, Queensland
  - Pfizer Investigational Site, Adelaide, South Australia
  - Pfizer Investigational Site, North Adelaide, South Australia
  - Pfizer Investigational Site, Prahran, Victoria
  - Pfizer Investigational Site, Subiaco, Western Australia

REFERENCES:
- [Derived] Marshall H, Nissen M, Richmond P, Shakib S, Jiang Q, Cooper D, Rill D, Baber J, Eiden J, Gruber WC, Jansen KU, Anderson AS, Zito ET, Girgenti D. Safety and immunogenicity of a booster dose of a 3-antigen Staphylococcus aureus vaccine (SA3Ag) in healthy adults: A randomized phase 1 study. J Infect. 2016 Nov;73(5):437-454. doi: 10.1016/j.jinf.2016.08.004. Epub 2016 Aug 9. PMID 27519620
- [Derived] Nissen M, Marshall H, Richmond P, Shakib S, Jiang Q, Cooper D, Rill D, Baber J, Eiden J, Gruber W, Jansen KU, Emini EA, Anderson AS, Zito ET, Girgenti D. A randomized phase I study of the safety and immunogenicity of three ascending dose levels of a 3-antigen Staphylococcus aureus vaccine (SA3Ag) in healthy adults. Vaccine. 2015 Apr 8;33(15):1846-54. doi: 10.1016/j.vaccine.2015.02.024. Epub 2015 Feb 21. PMID 25707693
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=6123K1-1007&StudyName=An%20Evaluation%20Of%20Three%20Dose%20Levels%20Of%203-Antigen%20Staphylococcus%20Aureus%20Vaccine%20%28SA3Ag%29%20In%20Healthy%20Adults